CLINICAL TRIAL: NCT01013909
Title: An Investigator-blind, Randomized, Multicenter, 5-arm, Placebo- and Active Controlled Parallel Group Pilot Trial to Explore the Efficacy and Tolerability of Topical Bifonazole Liquid Spray in Patients With Athlete's Foot.
Brief Title: Comparative Safety and Efficacy Study of New Bifonazol Spray vs Terbinafine Solution vs Placebo
Acronym: Porsche
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13957; 2008-005654-21 (EudraCT Number)
Record Dates: First submitted 2009-10-09; First posted 2009-11-16 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Tinea Pedis
Keywords: Bifonazole; Terbinafine; Reduced treatment duration; Efficacy; Safety; Athlete's foot; Moderate severity
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Drug: Bifonazole spray once daily
- Arm 2 (Experimental)
  Interventions: Drug: Bifonazole spray twice daily
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 5 (Active Comparator)
  Interventions: Drug: Lamisil Once

INTERVENTIONS:
Drug: Bifonazole spray once daily — Application of one dose daily by means of an metered dose
  Arms: Arm 1
Drug: Bifonazole spray twice daily — Application of two dose daily by means of an metered dose
  Arms: Arm 2
Drug: Placebo — Application of one dose daily by means of an metered dose
  Arms: Arm 3
Drug: Placebo — Application of one dose daily by means of an metered dose
  Arms: Arm 4
Drug: Lamisil Once — One application of Lamisil Once
  Arms: Arm 5

SUMMARY:
The study shall prove whether 6 consecutive doses of Bifonazole spray show comparable efficacy to a Terbinafine solution applied once.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 70 years
* Positive clinical findings of athlete's foot, limited to interdigital spaces, with a total athlete's foot severity score (AFSS) of at least 5 and not exceeding 10 points for the signs and symptoms of athlete's foot, and no sign or symptom scoring 'severe'

Exclusion Criteria:

* Clinical history suggestive of intolerance or allergies to one of the products or the ingredients of the products
* Plantar tinea pedis ("Mocassin-type")
* Onychomycosis of any toe
* Previous treatment with a systemic antifungal within 6 months prior to screening
* Previous treatment of feet with a topical antifungal within 4 weeks prior to screening
* Previous treatment with a topical antifungal applied to other areas of the body than feet within 2 weeks prior to screening
* Previous treatment of any topical medication applied to the feet within 2 weeks prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Assessment of erythema, scaling, vesiculation maceration, and pruritus based on a categorial scale (0=absent to 3 =severe), assessment of mycological cure based on cultures and microscopy | After 6 applications (7 and 42 days after start of treatment)
Local side effects on the skin | From day 1 through day 42

SECONDARY OUTCOMES:
Clinical cure | After 6 applications (7 and 42 days after start of treatment)
Mycological cure | After 6 applications (7 and 42 days after start of treatment)
Rate of negative culture | After 6 applications (7 and 42 days after start of treatment)
Rate of microscopy negative | After 6 applications (7 and 42 days after start of treatment)
Rate of absence of itching and burning | After 6 applications (7 and 42 days after start of treatment)
Incidence and severity of Adverse Event | From visit 2 (day 3) till visit 7 (day 42)
Vital Signs | Visit 1 (day 1) and visit 7 (day 42)
Local side effects | From visit 2 (day 3) till visit 7 (day 42)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here and search for websynopsis provided by the EMA — http://www.clinicaltrialsregister.eu